CLINICAL TRIAL: NCT06686225
Title: Comparative Effects of Bowen's Technique and Mulligan Bent Leg Raise Technique on Range of Motion and Function in Kabaddi Players With Hamstring Tightness
Brief Title: Bowens Technique Versus Mulligan Bent Leg Raise Technique in Kabaddi Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0432
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Sports Physical Therapy
Keywords: Endurance; Flexibility; Hamstring tightness; strength; sprinting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen's technique (Experimental): This group will receive 20 mint per session for 6 weeks of bowen's technique with moderate to high intensity of soft tissue mobilization.
  Interventions: Other: Bowen's technique.
- Bent leg raise technique. (Experimental): This group will receive 15 mints per session for 6 weeks of mulligan's bent leg raise technique with moderate to high intensity of soft tissue mobilization.
  Interventions: Other: Mulligan bent leg raise technique

INTERVENTIONS:
Other: Bowen's technique. — This group will receive 20 mint per session for 6 weeks of bowen's technique.
  * Frequency: 3-5 days per week for 6 days
  * Intensity: moderate to high intensity of soft tissue mobilization
  * Time: 20 mints
  * Type: Bowen's technique
  Arms: Bowen's technique
Other: Mulligan bent leg raise technique — This group will receive 15 mints per session for 6 weeks of mulligan's bent leg raise technique.
  * Frequency: 3-5 days per week for 6 days
  * Intensity: moderate to high intensity of soft tissue mobilization
  * Time: 15 mints
  * Type: Mulligan bent leg raise technique
  Arms: Bent leg raise technique.

SUMMARY:
The purpose of this study is to look into how Mulligan's bent leg raise technique and Bowen's technique affect the functional abilities and range of motion of hamstring-tight Kabaddi players. Our goal is to add to the expanding body of knowledge on sports rehabilitation by investigating the efficacy of various interventions and offering evidence-based suggestions for improving the health and performance of Kabaddi participants

DETAILED DESCRIPTION:
Few studies have been conducted to compare bowen's technique and Mulligan bent leg raise technique kabaddi players to enhance hamstring flexibility. Present study will seek to fill this gap by comparing the effects of Bowen's technique with mulligan bent leg raise technique in enhancing hamstring flexibility and functionality. Moreover, this study would ultimately aid coaches in designing effective training program for kabaddi players.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with hamstring tightness.
* Male
* Age between 18 to 30 years.
* 20° to 50° Active knee extension loss with hip in 90° of flexion.
* Full passive range of motion of knee extension (to rule out knee joint pathology)
* Subjects willing to participate in the study

Exclusion Criteria:

* Acute or chronic low back pain
* Subjects if they have any history of lower extremity injury in past 3 months
* Any fracture or surgery done for back, pelvis hip or knee.
* Any neurological symptoms involving prolapsed intervertebral disc or radiating pain.
* Spinal deformity
* Any recent abdominal surgery

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Active Knee Extension Test | 6 weeks
  The test measured the angle of the knee flexion with the help of a goniometer after the active knee extension with the hip stabilized at 90 degrees flexion. The angle of knee flexion represented the hamstring tightness. Each subject was positioned in supine position on the examination table. The lower limb which was not been examined was stabilized across the thigh with a strap. Another strap was used to stabilize the pelvis by placing the strap over the anterosuperior iliac spine. A line was drawn between the fibular head and the lateral malleolus. The angle of knee flexion of the subject was recorded from the goniometer in degrees.
Finger to Floor Test | 6 weeks
  The Finger to Floor Test was performed with the subject standing barefoot. The subject was asked to reach the floor with their finger-tips. The distance between the subject's long finger and the floor was measured using a standard measuring tape in centimeter's.
Sit and Reach Test | 6 weeks
  The test involved the subjects sitting on the floor with legs stretched out straight ahead. Footwear was removed and the soles of the feet were placed against the wall. Both the knees were locked and pressed flat on the floor. With the palm facing downward, the subject reached forward along the measuring line as far as he could ensure that the hands remain at the same level. The subject was asked to hold the end position for at least 2 seconds while the distance was being measured
Lower extremity functional scale | 6 weeks
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Arslan Aslam Malik, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zalleg D, Ben Dhahbi A, Dhahbi W, Sellami M, Padulo J, Souaifi M, Beslija T, Chamari K. Explosive Push-ups: From Popular Simple Exercises to Valid Tests for Upper-Body Power. J Strength Cond Res. 2020 Oct;34(10):2877-2885. doi: 10.1519/JSC.0000000000002774. PMID 30095736
- [Background] Malwanage KT, Senadheera VV, Dassanayake TL. Effect of balance training on footwork performance in badminton: An interventional study. PLoS One. 2022 Nov 17;17(11):e0277775. doi: 10.1371/journal.pone.0277775. eCollection 2022. PMID 36395192
- [Background] Pardiwala DN, Subbiah K, Rao N, Modi R. Badminton Injuries in Elite Athletes: A Review of Epidemiology and Biomechanics. Indian J Orthop. 2020 Mar 10;54(3):237-245. doi: 10.1007/s43465-020-00054-1. eCollection 2020 May. PMID 32399141
- [Background] Miranda-Oliveira P, Branco M, Fernandes O. Accuracy and Interpretation of the Acceleration from an Inertial Measurement Unit When Applied to the Sprint Performance of Track and Field Athletes. Sensors (Basel). 2023 Feb 4;23(4):1761. doi: 10.3390/s23041761. PMID 36850357
- [Background] Ikeda Y, Kijima K, Kawabata K, Fuchimoto T, Ito A. Relationship between side medicine-ball throw performance and physical ability for male and female athletes. Eur J Appl Physiol. 2007 Jan;99(1):47-55. doi: 10.1007/s00421-006-0316-4. Epub 2006 Oct 18. PMID 17047981
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Mehta SP, Fulton A, Quach C, Thistle M, Toledo C, Evans NA. Measurement Properties of the Lower Extremity Functional Scale: A Systematic Review. J Orthop Sports Phys Ther. 2016 Mar;46(3):200-16. doi: 10.2519/jospt.2016.6165. Epub 2016 Jan 26. PMID 26813750
- [Background] Adnan M, Arsh A, Ali B, Ahmad S. Effectiveness of bent leg raise technique and neurodynamics in patients with radiating low back pain. Pak J Med Sci. 2022 Jan-Feb;38(1):47-51. doi: 10.12669/pjms.38.1.4010. PMID 35035399
- [Background] Amjad F, Khalid A. Comparative effects of Bowen therapy and tennis ball technique on pain and functional disability in patients with thoracic myofascial pain syndrome. J Orthop Surg Res. 2023 Nov 24;18(1):895. doi: 10.1186/s13018-023-04379-z. PMID 37996838
- [Background] Javed S, Bashir MS, Mehmood A, Noor R, Ikram M, Hussain G. Comparative effects of post isometric relaxation technique and Bowen's therapy on pain, range of motion and function in patients with temporomandibular joint disorder. BMC Oral Health. 2024 Jun 12;24(1):679. doi: 10.1186/s12903-024-04440-1. PMID 38867195